CLINICAL TRIAL: NCT03705130
Title: Evaluation of Visual Performance With Contact Lenses
Status: Completed | Type: Observational
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Eric R. Ritchey, Assistant Professor, University of Houston
Other Study IDs: STUDY00000958
Record Dates: First submitted 2018-06-14; First posted 2018-10-15 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Myopia
Keywords: Multifocal Contact Lens; Myopia; Visual Performance
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group 1: All subjects will wear the 3 contact lenses: Single Vision, Multifocal 1 and Multifocal 2.
  Interventions: Device: Single Vision Contact Lens; Device: Multifocal Contact Lens 1; Device: Multifocal Contact Lens 2

INTERVENTIONS:
Device: Single Vision Contact Lens — Spherical Contact Lens worn on non-dispensing basis
  Other Names: comfilcon A
Device: Multifocal Contact Lens 1 — Multifocal Contact Lens worn on non-dispensing basis
  Other Names: comfilcon A
Device: Multifocal Contact Lens 2 — Multifocal Contact Lens worn on non-dispensing basis
  Other Names: etafilcon A

SUMMARY:
This study will evaluate the influence of contact lens optical design on visual performance using standard and multifocal soft contact lenses (MFCLs).

DETAILED DESCRIPTION:
The study will examine visual acuity with various contact lenses, with and without glare source, in myopes between the ages of 18-39 years old (inclusive) to determine the effect of different multifocal optical designs on visual performance in the post-fit period.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 39 years of age
* Best corrected visual acuity of at least 20/30
* Spherical equivalent refractive error in each eye of between -0.75 and -6.00 diopters sphere after vertexing to the corneal plane

Exclusion Criteria:

* Greater than -1.00 diopter of refractive astigmatism at the corneal plane
* Any active anterior segment disease, pathology, or surgery affecting vision, refraction, or the ability to wear a soft contact lens
* History of ocular trauma or surgery causing abnormal or distorted vision
* Current Rigid Gas Permeable (RGP) contact lens wearers
* Unwilling to have eyes photographed or video recorded
* Pregnant and/or lactating females, by self-report

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects between the ages of 18-39 (inclusive) without significant ocular disease.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Low Contrast Visual Acuity with Glare | Through study completion, an average of 3 hours
  Vision with contact lenses measured under low illumination conditions with glare source

SECONDARY OUTCOMES:
Low Contrast Visual Acuity without Glare | Through study completion, an average of 3 hours
  Vision with contact lenses measured under low illumination conditions without glare source

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nti AN, Gregory HR, Ritchey ER, Wolffsohn JS, Berntsen DA. Contrast Sensitivity with Center-distance Multifocal Soft Contact Lenses. Optom Vis Sci. 2022 Apr 1;99(4):342-349. doi: 10.1097/OPX.0000000000001874. PMID 35121719